CLINICAL TRIAL: NCT06261073
Title: Evaluation of Serum and Tissue Cathepsin L in Non-segmental Vitiligo Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Abdelrahim Abdelaal, Resident of dermatology ,venereology andandrology saqolta general hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-24-01-08MS
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with non-segmental vitiligo (Active Comparator): 30vitiligo patients their age above 18 years attending dermatology outpatient clinics of Sohag University hospital.
  Interventions: Diagnostic Test: blood sample and tissue biopsy
- healthy volunteers. (Active Comparator): .A group of age and sex- matched healthy participants will be included as a control group.
  Interventions: Diagnostic Test: blood sample and tissue biopsy

INTERVENTIONS:
Diagnostic Test: blood sample and tissue biopsy — Serum level of Cathepsin L: 3 cm of blood will be taken on EDTA tubes from patients and control subjects and will be analyzed by double antibody sandwich enzyme-linked immune-sorbent assay (ELISA) to assess the level of CTSL in blood samples. Tissue expression of Cathepsin L: 5 mm punch biopsies will be taken under local anesthesia from lesions and from the adjacent normal skin of patients (from the lesional and peri-lesional sites). Also, skin biopsy of normal skin will be taken from healthy volunteers. The specimen of skin will be immediately placed in a formalin saline, and then immune-histochemical evaluation will be done to evaluate the CTSL expression in tissue.

SUMMARY:
Introduction Vitiligo is an autoimmune disease of the skin that targets pigment producing melanocytes and results in patches of depigmentation that are visible as white spots (Frisoli et al., 2020) Vitiligo is a relatively common acquired pigmentation disorder that can cause significant psychological stress (Leung AKC et al., 2021). The disease affects both genders equally, it can appear at any age, and the average age of onset is somewhat variable in different geographic (Majumder et al, 1993), with an estimated prevalence of 0.5-2% of the population in both adults and children worldwide (Krüger et al, 2012).

Vitiligo results in white macules and patches on the body. Initial lesions occur most frequently on the hands, forearms, feet, and face, favoring a periocular or perioral distribution (Ahmed jan N et al., 2023). Vitiligo lesions are classified into 2 major categories: segmental vitiligo (SV) and non-segmental vitiligo (NSV) (Relke et al ., 2019). Segmental vitiligo is characterized by its early onset, rapid stabilization, and unilateral distribution (Van Geel et al., 2017). Non-segmental vitiligo comprises of generalized (vitiligo vulgaris), acrofacial, mucosal (multifocal), and universal vitiligo (Kovacevic et al., 2016). Non-segmental vitiligo (NSV) is the most common form of vitiligo (Benzekri et al., 2013). Multiple mechanisms are involved in melanocyte disappearance, namely genetic predisposition, environmental triggers, metabolic abnormalities, impaired renewal, and altered inflammatory and immune responses (Boniface K et al ., 2018).

The results of some studies indicate a frequent association of vitiligo with autoimmune diseases. A number of studies have established a higher prevalence of autoimmune endocrine diseases in women, as well as in non-segmental vitiligo patients and in cases of family history of vitiligo and/or other autoimmune diseases. In addition, it was shown that the prevalence of endocrine diseases increases with increasing area of depigmentation (Troshina EA et al., 2020). Autoimmunity in vitiligo is driven by the IFN-γ-CXCL10 cytokine signaling pathway. Activated melanocyte-specific CD8+ T cells secrete IFN-γ, which signals through the IFN-γ receptor (IFN-γR) to activate JAK1/2 and STAT1. This induces the production of CXCL9 and CXCL10, which signal through their receptor CXCR3 to recruit more auto-reactive T cells to the epidermis, resulting in widespread melanocyte destruction (Harris JE et al., 2017).

The lysosomal cysteine proteinases of the papain family are involved in lysosomal bulk proteolysis, major histocompatibility complex class II-mediated antigen presentation, pro-hormone processing, and extracellular matrix remodeling.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-segmental vitiligo attending the dermatology outpatient clinics of Sohag University hospital. A group of age and sex- matched healthy participants will be included as a control group.

Exclusion Criteria:

* (A) Pregnancy and lactation. (B) Patients on topical and systemic treatment for vitiligo in the last 4weeks prior to enrollment in the study.

(C) Malignacies. (D) Patients with systemic diseases, diabetes, hypertension and bleeding disorders.

(E) Patients who are receiving chemotherapy or radio therapy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Cathepsin L | 12 months
  3 cm of blood will be taken on EDTA tubes from patients and control subjects : 5 mm punch biopsies will be taken under local anesthesia from lesions and from the adjacent normal skin of patients

REFERENCES:
- [Background] Ghasemi M, Bajouri A, Shafiiyan S, Aghdami N. Hair Follicle as a Source of Pigment-Producing Cells for Treatment of Vitiligo: An Alternative to Epidermis? Tissue Eng Regen Med. 2020 Dec;17(6):815-827. doi: 10.1007/s13770-020-00284-2. Epub 2020 Oct 9. PMID 33034877
- [Background] Kageshita T, Yoshii A, Kimura T, Maruo K, Ono T, Himeno M, Nishimura Y. Biochemical and immunohistochemical analysis of cathepsins B, H, L and D in human melanocytic tumours. Arch Dermatol Res. 1995;287(3-4):266-72. doi: 10.1007/BF01105077. PMID 7598531
- [Background] Kawada A, Hara K, Kominami E, Hiruma M, Noguchi H, Ishibashi A. Processing of cathepsins L, B and D in psoriatic epidermis. Arch Dermatol Res. 1997 Jan;289(2):87-93. doi: 10.1007/s004030050160. PMID 9049042
- [Background] Kovacevic M, Stanimirovic A, Vucic M, Goren A, Situm M, Lukinovic Skudar V, Lotti T. Mixed vitiligo of Blaschko lines: a newly discovered presentation of vitiligo responsive to combination treatment. Dermatol Ther. 2016 Jul;29(4):240-3. doi: 10.1111/dth.12345. Epub 2016 Mar 11. PMID 26970077